CLINICAL TRIAL: NCT04726020
Title: NICSO National Study: Physician - Nurse Monitoring Project About Oncological Adverse Events
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NICSO
Record Dates: First submitted 2020-09-08; First posted 2021-01-27 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Cancer
Keywords: immunotherapy; targeted therapy; chemotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Two comparison groups: an intervention group (intensive phone monitoring of adverse event reactions) compared with a placebo group (standard monitoring)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive monitoring (Experimental): Intensive phone monitoring of drug adverse events
  Interventions: Other: Intensive monitoring
- Standard monitoring (Placebo Comparator): Standard monitoring of drug adverse events
  Interventions: Other: Standard monitoring

INTERVENTIONS:
Other: Intensive monitoring — periodic and planned monitoring nurse intervention with phone call
  Arms: Intensive monitoring
Other: Standard monitoring — standard monitoring of adverse event reaction
  Arms: Standard monitoring

SUMMARY:
The lacking adherence to guidelines on prevention and treatment of different chemotherapy, targeted therapy, and immunotherapy induced toxicities is the reason why there are a potential incidence and duration increase of adverse events. It is clear the need of a collateral effect early recognition for an adequate clinical management and for limiting their intensity and duration.

There is the need for a multicentre randomized clinical study in specific therapeutical settings (chemotherapy, target therapy, immunotherapy) assessing the impact of planned and ongoing patients' monitoring by nurses.

The NICSO study foresees patient enrolment that is in adjuvant chemotherapy for breast cancer, colon, and lung; that is in chemotherapy or immunotherapy or with targeted therapy. Moreover, this working assesses toxicity differences (but also of QoL, number of PS access or non-planned medical examinations, number of hospitalization and number of recovery days) in patients that carried out a toxicity prevention and cure standard therapy in comparison with the standard assessment to which is added a periodic nursing phone intervention.

DETAILED DESCRIPTION:
The lacking adherence to guidelines on prevention and treatment of different chemotherapy, targeted therapy, and immunotherapy induced toxicities is the reason why there are a potential incidence and duration increase of adverse events. It is clear the need of a collateral effect early recognition for an adequate clinical management and for limiting their intensity and duration.

A better toxicity management can have a positive impact on a correct treatments dose-intensity. Scientific community debate on toxicity assessment ways and means is still open. The most debated questions concern:

* Physician and/or patient reporting adverse events;
* Nurse role in the adverse events assessment;
* How much assessment methods (assessment frequency, who's involved in adverse events monitoring) means for:

  * Time spent with toxicity and intensity reduction;
  * Treatment adherence. Some literature evidence is avaiable and support the need of intensive monitoring of patients in terms of adverse events. However, there is the need for a multicentre randomized clinical study in specific therapeutical settings (chemotherapy, target therapy, immunotherapy) assessing the impact of planned and ongoing patients' monitoring by nurses.

This is a multi-centric, randomized, open comparative study design, between a planned and consecutive monitoring nurse intervention in addition to the chemotherapy toxicity prevention and cure standard therapy package insert (chemotherapy, target therapy, immunotherapy), and the only use of the cancer therapy toxicity prevention and cure standard therapy package insert (chemotherapy, target therapy, immunotherapy).

The study involves All the patients with a solid tumor on treatment with adjuvant chemotherapy or receiving target therapy or immunotherapy for the first time in their cancer history.

This study design will last 24 months. Patient recruitment will last 18 months from the beginning of the study. The study period will be 4 months for the group on treatment with immunotherapy and target therapy and at least 6 months for the group on treatment with adjuvant chemotherapy. The study could be interrupted when there is a therapy withdrawal because of cancer progression, severe toxicity or for the informed consent for withdrawal, or because of death. If there is a temporary interruption or a treatment withdrawal period, patients still are in under monitoring, according to their group. The study will end with the end of the planned period monitoring, which is the last call to the enlisted patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18;
* Solid cancer histological diagnosis on treatment with one of the listed medicines, defined by treatment type:

  * Adjuvant chemotherapy:

    * anthracyclines and cyclophosphamide ± taxanes (breast cancer)
    * oxaliplatin e fluoropyrimidine (colon cancer)
    * combination of platin or its derivate (lung cancer)
  * First line oral target therapy:

    * sunitinib, pazopanib (renal cancer)
    * gefitinib, erlotinib,afatinib, crizotinib (lung cancer)
    * vemurafenib ± comimetinib, dabrafenib±trametinib (Melanoma)
    * everolimus ± exemestane (breast cancer)
    * vandetanib o lenvatinib (thyroid cancer)
    * vismodegib (skin basal cell carcinoma)
    * imatinib (GIST)
  * Immunotherapy:

    * drugs anti CTLA4
    * drugs antiPD1/PDL-1
    * their combination
    * sign of informed consent form;
    * phone call availability and accessibility;
    * life expectancy higher than 6 months.

Exclusion Criteria:

* Presence of cerebral symptomatic metastasis;
* Presence of neurological or psychiatric disease or other conditions that stop the protocol procedure compliance;
* Previous systemic cancer treatment. These exclusion criteria are justified because usually a systemic cancer treatment cause changes in toxicity profile. This means that these patients have higher attention on their toxicities and probably receive codified preventive treatments already.
* Participation in other clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 645 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Assessment of the number of days that have passed with at least a toxicity grade >= 3 | 6 months
  Assessment of the number of days that have passed with at least a toxicity grade >= 3. The assessed toxicities have been chosen for their clinical relevance and for their higher danger to reduce patients' treatment adherence, invalidating therapy benefits.

SECONDARY OUTCOMES:
low grade toxicity (grade 1 and 2) incidence and duration | 6 months
  incidence and duration of grade 1 and 2 toxicity
number of ER admissions and number of non-planned medical examinations | 6 months
  number of ER admissions and number of non-planned medical examinations
number of hospitalization and its duration because of treatment toxicity | 6 months
  number of hospitalization and its duration because of treatment toxicity
QoL (Quality of Life) assessment | 6 months
  administration of validated questionnaires and evaluation of patients'quality of life

OTHER OUTCOMES:
Changes in treatment dose intensity | 6 months
  Changes intreatment dose intensity (Dose intensity)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bossi, MD, Study Chair — Italian Network of Supportive Care in Cancer; Andrea Antonuzzo, MD, Study Chair — Italian Network of Supportive Care in Cancer
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

DOCUMENTS (1):
  • Study Protocol (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/20/NCT04726020/Prot_000.pdf